CLINICAL TRIAL: NCT05245812
Title: Safety and Feasibility of Robotic Single-port (SP) Nipple Sparing Mastectomy: A Single Institution, Single Arm Pilot Trial
Brief Title: Safety and Feasibility of Robotic SP Nipple Sparing Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deborah Farr, MD (Other)
Responsible Party: Sponsor-Investigator, Deborah Farr, MD, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2022-0091
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; High Risk of Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment arm (SPrNSM) (Experimental): Patients will undergo Single Port robotic Nipple Sparing Mastectomy (SPrNSM) with immediate breast reconstruction with tissue expanders/implants and acellular dermal matrix (Alloderm)
  Interventions: Device: da Vinci SP Surgical System

INTERVENTIONS:
Device: da Vinci SP Surgical System — This is a software-controlled, electro- mechanical system designed for surgeons to perform single port minimally invasive surgery.
  Other Names: da Vinci SP Surgical System, Model SP1098

SUMMARY:
This is a single arm, single-center, prospective clinical trial designed to track the peri, post-operative and oncologic outcomes when utilizing the da-Vinci single port (SP) robotic platform to perform robotic nipple sparing mastectomy (rNSM) and immediate breast reconstruction with tissue expanders/implants and acellular dermal matrix (ADM - Alloderm), for patients with breast cancer as well as those with a high risk for breast cancer.

Safety and feasibility measures will be measured as primary outcome measures. Oncological and patient satisfaction outcome measures will be measured. Our hypothesis is that SPr-NSM is equal to open NSM in terms of safety, feasibility and oncological outcomes with improved patient satisfaction as measured by nipple sensation and patient reported outcomes.

DETAILED DESCRIPTION:
rNSM using the multi-port robotic platform followed by standard of care open breast reconstruction has been done successfully at multiple institutions worldwide with comparable, if not superior outcomes to an open surgical approach. This study explores this procedure with the Da Vinci SP robot with pre-pectoral reconstruction with acellular dermal matrix. The patients will be evaluated per standard of care post-operative visits at 2 weeks, 1 month, and every 6 months for five years post operatively for subjective patient satisfaction and objectively for post-operative nipple sensation. The patients will be monitored longitudinally for oncologic outcomes including the presence of a new breast cancer and/or breast cancer recurrence. Patients will be monitored for any complications related to rNSM and the use of ADM in expander and implant-based breast reconstruction.

Investigational Device:

The da Vinci SP Surgical System, Model SP1098 is a software-controlled, electro- mechanical system designed for surgeons to perform single port minimally invasive surgery. The Model SP1098 Surgical System consists of a Surgeon Console, a Patient Cart, and a Vision Cart, and is used with a Camera Instrument, EndoWrist SP Instruments, and Accessories.

Indications for Use:

The da Vinci SP Surgical System, Model SP1098 is cleared for use in urologic surgical procedures that are appropriate for a single-port approach and transoral otolaryngology procedures restricted to T1 and T2 tumors. This investigational study will evaluate device usage in nipple sparing mastectomy (NSM) procedures.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for open nipple sparing mastectomy, per standard of care with regards to anatomic factors and tumor location including: nipple sparing resection and resection OR prophylactic mastectomy for risk reduction OR treatment of ductal carcinoma in-situ or clinically node negative cT1-T3 breast cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Inability to provide informed consent
* Pregnant or nursing women
* Patients with:
* Inflammatory breast cancer
* Skin involvement with tumor
* Pre-operative diagnosis of Nipple Areolar Complex (NAC) tumor involvement
* Grade 3 or higher nipple ptosis
* Contraindicated for general anesthesia or surgery
* Heavy current smoking history (defined as > 20 cigarettes per day)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete single port nipple sparing mastectomy (SPrNSM) | Date of surgery (Day 1)
  The number of participants who complete single port nipple sparing mastectomy (SPrNSM) will be measured.
Incidence of perioperative complications | 30 days following surgery
  Perioperative complications will be described using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTACAE) v. 4.03 criteria. Complications will refer to any medical occurrence directly attributed to the surgical procedure during and within the first 30 days following use of the SP robotic platform and ADM. Grade 3, 4, or 5 complication or adverse event will constitute an event. Perioperative complication rates will be compared to historical complication rates.

SECONDARY OUTCOMES:
Number of participants with positive margins | 2 weeks following date of surgery
  The pathologist will assess margin status in patients undergoing SPrNSM
Number of participants with new breast cancers | following date of surgery up to 5 years
  The PI will assess new breast cancers.
Number of participants with recurrent breast cancers | following date of surgery up to 5 years
  The PI will assess recurrent breast cancers.
Patient satisfaction as measured by BREAST-Q reconstruction tool | Baseline, postoperatively at 2 weeks, every 6 months for 5 years
  Patient satisfaction is measured by BREAST-Q reconstruction tool at baseline, postoperatively at 2 weeks, and every 6 months for 5 years. BREAST-Q reconstruction module and Breast implant illness survey for patients. Questions about self-confidence, comfort, acceptance of new appearance, feeling of implants, breast pain. The score represents questionnaires about different domains and each question has four possible dimensions. The values of these dimensions varies from 1 (minimum score- worst outcome) to 4 or 5 (maximum score- best outcome) (Likert Scale) depending on part of the questionnaire .
Patient satisfaction as measured by BREAST-Q sensation tool | Baseline, postoperatively at 2 weeks, every 6 months for 5 years
  Patient satisfaction is measured by BREAST-Q sensation tool at baseline, postoperatively at 2 weeks, and every 6 months for 5 years and it is another tool to help quantify breast sensation both pre-operatively and post-operatively. The Breast-Q is comprised of 2 domains - i) Satisfaction domains and ii) Well-being domains, which are further divided into sub-domains. We will be using 3 satisfaction sub-domains: i) Satisfaction with breasts ii) Satisfaction with Nipple iii) Satisfaction with outcome and 3 well-being sub-domains: i) Psychosocial well-being ii) Sexual well-being and iii) Physical well-being. The values range from 1 (minimum score- worst outcome) to 4 or 5 (maximum score- best outcome) (Likert Scale) depending on part of the questionnaire.
Degree to which the patients maintain nipple sensation as measured by Semmes Weinstein monofilament tool at baseline | Baseline, postoperatively at 2 weeks, every 6 months for 5 years
  Degree to which the patients maintain nipple sensation will be measured by Semmes Weinstein monofilament tool at baseline, postoperatively at 2 weeks, and every 6 months for 5 years. Monofilament diameter and force will be measured at 9 different locations of the breast to determine the degree of sensation.
Incidence of short term complications | Post-operatively at 30 days
  Reconstruction outcomes is measured by short term complications (wounds, infections, seromas, and device exchange or loss) that occur post-operatively after surgery Short term complications will be described using the NCI CTACAE v. 4.03 criteria.
Incidence of long term complications | Following surgery up to 5 years
  Long term complications will be described using the NCI CTACAE v. 4.03 criteria and will refer to any medical occurrence directly attributed to the surgical procedure up to 5 years following use of the SP robotic platform and ADM. Grade 3, 4, or 5 complication or adverse event will constitute an event.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Farr, MD, FACS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farr DE, Haddock NT, Tellez J, Radi I, Alterio R, Sayers B, Zeh H 3rd. Safety and Feasibility of Single-Port Robotic-Assisted Nipple-Sparing Mastectomy. JAMA Surg. 2024 Mar 1;159(3):269-276. doi: 10.1001/jamasurg.2023.6999. PMID 38231502